CLINICAL TRIAL: NCT02244580
Title: Evaluation of the MammaTyperTM Kit, Ref 90020/90021 Performed on Clinical Material Obtained From Patients With Breast Cancer: Re-Examination of Tumor Material and Re-Evaluation of Patient Data of the FinHer-Study
Brief Title: Re-Evaluation of Tumor Samples From Women With Breast Cancer With the in Vitro Diagnostic Kit "MammaTyperTM"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioNTech Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MammaTyper-FinHer
Record Dates: First submitted 2014-09-04; First posted 2014-09-19 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Invasive Breast Cancer
Keywords: Subtyping of Invasive breast cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MammaTyper™ (Experimental): MammaTyper™ kit will be used tio assess tumor material of patients enrolled into the FinHer trial.
  Interventions: Device: MammaTyper™

INTERVENTIONS:
Device: MammaTyper™ — MammaTyper™ kit is a molecular in vitro diagnostic test for the quantitative detection of the ribonuclease acid (RNA) expression status of the genes for estrogen receptor (ESR1), progesterone receptor (PGR), human epidermal growth factor receptor 2 (HER2) and proliferation antigen KI 67.

SUMMARY:
This is a prospective examination of tumor material of breast cancer patients randomized into the FinHer-trial (= (= Comparison of vinorelbine and docetaxel and trastuzumab as adjuvant treatments of breast cancer patients wirh a high risk of cancer recurrence).

The formalin-fixed, paraffin-embedded tissue samples will be analysed for Estrogen receptor 1 (ESR1), progesterone receptor (PgR), Human epidermal growth factor receptor 2 (HER2) and Antigen Ki-67 (Ki-67) with the molecular in vitro diagnostic kit MammaTyper™.

According to the new subtyping the 5 year Distant disease free survival (DDFS) and Overall survival (OS) will be re-evaluated.

DETAILED DESCRIPTION:
Despite the fact that reliable measures for the markers ESR1, PgR, HER2, Ki-67 are necessary with the currently used methods up to 20% of determinations are inaccurate and especially Ki67- measures are not very reproducible. Therefore new evaluation systems or new methods are necessary to improve diagnostic.

At least 4 subtypes can be distinguished to date depending on the expression of ESR, PgR, Her2 and Ki-67:

* Luminal A-type
* Luminal B-type
* Her2-type
* Triple-negative-type

MammaTyper™ uses a new approach. Instead of detection of the marker proteins, the messenger ribonucleic adic (mRNA) of marker proteins is quantitated. This prospectively planned diagnostic study will investigate the potential of subgrouping of patients at baseline according to results of MammaTyper™ methodology for predicting survival.

Patients will be subgrouped according to the new marker determination and the DDFS and OS will be evaluated and compared to the DDFS and OS of subgrouping with former marker determination.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer verified in a histological biopsy
* Age 65 or younger
* Estrogen receptor (ER), PgR and HER2 expression have been determined
* No distant metastases present (M0)
* The patient provides a written informed consent for study participation
* The estimated risk of breast cancer recurrence is high (25% or higher within the first 5 years from the date of the diagnosis, over >35% within the first 10 years from the diagnosis)

Exclusion Criteria:

* Patients with breast cancer with "a special histological type" (mucinous, papillary, medullary, or tubular type of breast cancer) when no metastases are present in the ipsilateral axillary lymph nodes
* The WHO performance status is moderate/poor, Z >1
* The peripheral blood leukocyte count is less than 3.0 x 109/L, the blood granulocyte count is less than 1.5 x 109/L, or the blood thrombocyte count is less than 120 x 109/L
* Any physical or mental disorder that is considered to prohibit administration of chemotherapy
* Cardiac failure; severe cardiac arrythmia requiring regular medication

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2014-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Oed, Dr., Study Director — BioNTech Diagnostics GmbH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical data and breast tumour tissue samples were collected within the FinHer trial (identifier ISRCTN76560285), where 1010 women with axillary node-positive or high-risk axillary node-negative breast cancer were randomly assigned between October 2000 and September 2003.
Groups:
- MammaTyper™: MammaTyper™ kit will be used to assess tumor material of patients enrolled into the FinHer trial.
  MammaTyper™: MammaTyper™ kit is a molecular in vitro diagnostic test for the quantitative detection of the ribonuclease acid (RNA) expression status of the genes for estrogen receptor (ESR1), progesterone receptor (PGR), human epidermal growth factor receptor 2 (HER2) and proliferation antigen KI 67.
Period: Overall Study
Arm/Group | MammaTyper™
Started | 1010
Completed | 769 (An RT-qPCR assay was performed from breast cancer tissues of 769 out of the 1010 patients.)
Not Completed | 241
Not completed — No cancer tissues available | 241

BASELINE CHARACTERISTICS:
Population: Clinical data and breast tumour tissue samples were collected within the FinHer trial (identifier ISRCTN76560285).
Groups:
- FinHer Patients: Of all patients, FFPE tumour block was processed with the RNXtract RNA extraction kit (BioNTech Diagnostics GmbH, Mainz) using a magnetic particle-based assay (Supplemental file 1A).
  RT-qPCR was done with the MammaTyper kit (BioNTech Diagnostics GmbH, Mainz) for ESR1, PGR, ERBB2 and MKI67.
Arm/Group | FinHer Patients
Number analyzed (Participants) | 1010
Age, Continuous [Median (Full Range); unit: years] | 50.9 [25.5 to 65.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1010
  Male | 0
Region of Enrollment [Number; unit: participants]
  Finland | 1010

OUTCOME MEASURES:

1. Primary Outcome: 5 Year Distant Disease Free Survival (DDFS) Assessed as Rate of Patients Without Distant Metastases in Subgroup Luminal A vs. Combined Subgroup (Luminal B, HER2 Positive, Triple Negative), Based on Subtyping With MammaTyper™
Description: Tumor material of breast cancer patients will be newly assessed by MammaTyper™ and 5 year DDFS will be calculated new according to new subgrouping (Luminal A vs. combined subgroup (Luminal B, HER2 positive, triple negative))
Time Frame: 5 year from the date of patient randomisation
Measure: Number; unit: percentage of analyzed participants
Groups:
- Luminal A: Patients subtyped as Luminal A with DDFS determined 5 years after randomisation
- Combined Subtype: Patients subtyped as Luminal B, HER2 positive, triple negative with DDFS determined 5 years after randomisation
Arm/Group | Luminal A | Combined Subtype
Number analyzed (Participants) | 769 | 769
percentage of analyzed participants | 92 | 82
Statistical Analysis 1: Comparison: Luminal A vs Combined Subtype; Test type: Superiority or Other; p = 0.0018, Regression, Cox; Hazard Ratio (HR) = 0.423, 95% CI 2-sided [0.246 to 0.726]

2. Secondary Outcome: Number of Patients With High Ki-67 and Prognosis on Outcome for DDFS and OS (Measured by Hazard Ratio)
Description: High Ki-67 is prognostic for worse outcome for DDFS and OS (measured by hazard ratio)
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Groups:
- Patients With MKI67 mRNA Determination: Patients with low MKI67 mRNA
Arm/Group | Patients With MKI67 mRNA Determination
Number analyzed (Participants) | 769
Hazard ratio | 0.42 [0.25 to 0.71]
Statistical Analysis 1: Comparison: Patients With MKI67 mRNA Determination; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.25 to 0.71]

3. Secondary Outcome: Number of Patients With Ki-67 Determined by MammaTyper™ Compared to Local Ki-67 Eyeballed Assessment for Luminal Tumors and Correlation to Rate of Patients With Regard to OS and DDFS
Description: Superiority of outcome prediction for MammaTyper™ Ki-67 over local Ki-67 eyeballed assessment for Luminal tumors with regard to OS and DDFS
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Hazard ratio
Groups:
- DDFS According to MKI67 mRNA and Ki-67 Protein (IHC) Levels: Determination of DDFS of patients according to MKI67 mRNA (RT-qPCR) and Ki-67 protein (IHC) levels
- OS According to MKI67 mRNA and Ki-67 Protein (IHC) Levels: Determination of OS of patients according to MKI67 mRNA (RT-qPCR) and Ki-67 protein (IHC) levels
Arm/Group | DDFS According to MKI67 mRNA and Ki-67 Protein (IHC) Levels | OS According to MKI67 mRNA and Ki-67 Protein (IHC) Levels
Number analyzed (Participants) | 769 | 769
Hazard ratio
  DDFS (MKI67 mRNA positive - negative) | 0.42 [0.25 to 0.71] | 0.45 [0.23 to 0.88]
  DDFS (Ki-67 protein positive - negative) | 0.56 [0.37 to 0.84] | 0.43 [0.24 to 0.77]

ADVERSE EVENTS:
Groups:
- EG000: Since only tumor material was used, adverse events were not documented within the MammaTyper Study
Arm/Group | EG000
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No